CLINICAL TRIAL: NCT01659814
Title: Dopamine Neurotransmission in Major Depression
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Diego A. Pizzagalli, Associate Professor, Department of Psychiatry, Harvard Medical School, Mclean Hospital
Other Study IDs: 2009P000038
Record Dates: First submitted 2012-08-02; First posted 2012-08-08 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Major Depressive Disorder; Anhedonia
Keywords: Major Depressive Disorder; Anhedonia; Dopamine; Electroencephalography (EEG); Positron Emission Tomography (PET); Reward
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Individuals with Major Depressive Disorder
- Healthy Control Individuals

SUMMARY:
The overall aim of this study is to utilize an integrative research model in order to dynamically assess reward-related dopamine (DA) transmission in major depressive disorder (MDD) and test the role of dysfunctional DA release in depression and anhedonia.

The first arm of this line of research (PET scan) aims to investigate phasic DA release in MDD during incentive motivation. The investigators will utilize an established molecular imaging technique to measure striatal DA release dynamically during performance of testing and control versions of a monetary incentive delay task, which involves anticipation and receipt of monetary rewards. In doing so, this experiment will link together independent lines of research that have associated depression with decreased hedonic responsiveness, impaired reinforcement learning and dysfunctional DA transmission. We hypothesize that, relative to matched controls, unmedicated MDD subjects will show reduced reward-related ligand (11C-raclopride) displacement. Reduced ligand displacement will be interpreted as indicating reduced task-induced release of endogenous striatal DA in response to reward-predicting cues and unpredictable reward in MDD subjects.

In the second arm of this research (EEG recording), the investigators aim to probe the spatio-temporal dynamics of brain mechanisms underlying positive and negative reinforcement learning in MDD and their relations to phasic DA. Participants will perform the probabilistic stimulus selection task (PSST) while event-related potentials (ERPs) are collected. The investigators expect that, relative to matched controls, unmedicated MDD subjects will show reduced positive reinforcement learning, potentiated negative reinforcement learning, and larger (i.e., more negative) feedback-related negativity (FRN) in response to positive reinforcement (indicative of reduced DA transmission). Moreover, the investigators hypothesize that a more negative FRN in response to positive reinforcement will be associated with decreased striatal raclopride displacement (i.e., lower release of endogenous DA) as measured by PET in the first part of the study. This experiment will investigate the effects of blunted DA transmission on behavioral and ERP markers of both positive and negative reinforcement learning.

ELIGIBILITY:
Inclusion Criteria:

* Both genders and all ethnic origins, age between 18 and 45;
* Written informed consent;
* Right-handed (Chapman and Chapman 1987);
* Absence of serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease;
* Absence of history of seizure disorder;
* Absence of history of current diagnosis of any of the following DSM-IV psychiatric illnesses: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, substance dependence, substance abuse within the last 12 months (with the exception of cocaine or stimulant abuse; which will lead to exclusion), as assessed by subject history and a structured clinical interview (SCID-I/NP);
* Absence of history of cocaine or stimulant use (e.g., amphetamine, cocaine, methamphetamine);
* Absence of history of use of dopaminergic drugs (including methylphenidate);
* Absence of current use of other psychotropic drugs
* Absence of substance dependence or substance abuse in the last 12 months;
* Absence of history or current diagnosis of dementia, or a score greater than 26 on the Mini Mental Status Examination (Folstein, 1975) at the screening visit;
* Absence of clinical or laboratory evidence of hypothyroidism;
* Absence of neurological illness

Specific exclusion criteria for PET scan are as follows:

* Pregnant women, women trying to get pregnant, or women of childbearing potential who are not using a medically accepted means of contraception (defined as implant, condom, diaphragm, spermicide, IUD, s/p tubal ligation, partner with vasectomy).
* Failure to meet standard PET safety requirements.

Specific inclusion criteria for depressed participants are as follows:

* DSM-IV diagnostic criteria for MDD melancholia subtype (diagnosed with the use of the SCID) or MDD with anhedonia (score of 3 or greater on the Snaith-Hamilton Pleasure Scale (SHPS));
* A baseline HRSD score (Hamilton 1960) greater than or equal to 16 (17-item version);
* Absence of suicidal ideation where outpatient treatment is determined unsafe by the study clinician. These patients will be immediately referred to appropriate clinical treatment;
* Absence of past or current mood congruent or incongruent psychotic features;
* Absence of lifetime history of electroconvulsive therapy (ECT)
* Subjects taking antidepressants at the time of their screening visit will be enrolled only if they are willing (after discussing with their prescribing clinician), and the study clinician determines that it is clinically appropriate for them to discontinue their current antidepressant for a period greater than five half-lives of their current medication (but no longer than 7 days). For these subjects, the baseline visit and the first physiology session will only occur after the 7 day interval has passed.

Specific inclusion criteria for control participants are as follows:

* Absence of any psychiatric illness (including alcohol and substance abuse), as assessed by subject history and a structured clinical interview (SCID-I/NP).
* Absence of any medication for at least three weeks.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with Major Depressive Disorder and Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Event-Related Potentials (ERPs) during PSST task | At session 3, during the EEG recording
  ERPs will be generated during performance of the probabilistic stimulus selection task (PSST). Feedback-locked ERPs will be computed within epochs starting 100 ms before the feedback and lasting 924 ms. ERPs will be baseline-corrected to the first 100 ms of the extracted epoch. The feedback-related negativity (FRN) will be defined as the most negative peak 200-400 ms at frontocentral electrodes (Fz, FCz, Cz) after positive or negative feedback.
  Group (MDD vs. controls) x Trial Type (accuracy on Choose A vs. Avoid B) mixed ANOVA will be performed to test the hypothesis that relative to controls, MDD subjects will show reduced positive reinforcement learning but potentiated negative reinforcement learning. Group x Feedback Type (positive vs. negative) mixed ANOVA will be performed to test the hypothesis that MDD subjects will show larger FRN in response to positive reinforcement.
[11C]raclopride binding potential | At session 2, during the PET scan
  [11C]Raclopride binding potential will be recording during participant's performance of the monetary incentive delay (MID) task and is taken as an indication of release of endogenous dopamine. A reduction in raclopride binding potential is taken as an indication of increased extra-cellular dopamine concentration.
  A reference tissue method will be used to calculate voxelwise binding potential and generate statistical parametric images of changes in binding potential. The cerebellum will be used as reference tissue. In addition to voxelwise analyses, a regions-of-interest approach will be used to extract binding potential from caudate nucleus, putamen and ventral striatum using the procedure described by Laruelle's group. A multivariate analysis of variance (MANOVA) considering various striatal regions and using Group (MDD vs. Controls) as between-subject factor and Condition (reward vs. control task) as repeated measure will be performed.

SECONDARY OUTCOMES:
Behavioral Performance in Monetary Incentive Delay task | During session 2
  Data recorded include response time and accuracy.
  The task was modeled after prior work in non-human primates in order to maximize our ability to detect changes in [11C]raclopride binding potential, which will be taken as an indication of release of endogenous dopamine. At the outset of each trial, a visual cue signaling either potentially rewarding outcomes or no monetary incentive will be presented. After a fixed interval, participants will press a button in response to a red square target. A second interval will follow the target, after which visual feedback will notify participants whether they have won or not won money.
  In the reward version of the task, 150 trials will be presented over 25 min. Among these trials, 112 will be reward and 38 will be no-incentive trials. For successful trials, based on participant's response time, participants earn between $1.00 and $1.80.
Behavioral Performance in Probabilistic Stimulus Selection Task (PSST) | During session 3
  Data recorded include response time and accuracy.
  The PSST task examines whether participants exhibit a bias for choosing frequently reinforced stimuli or avoiding frequently punished stimuli, and thus to assess positive and negative reinforcement learning. MDD subjects and individuals at increased risk for depression are expected to be better at learning from punishment than reward in the PSST.
  The task has two phases: a learning and a testing phase. In the learning phase, subjects are randomly presented with three different stimuli pairs (AB, CD, EF), and are instructed to choose one of the two stimuli by pressing a key. After the response, feedback is given to indicate whether the choice was correct or incorrect. Feedback is probabilistic and one stimulus in each pair is correct more often than the other.
Questionnaire Data | Sessions 1-3
  Throughout the study, participants will complete self-report questionnaires assessing mood, stress levels, hedonic state, caffeine intake, nicotine intake and craving, and alcohol intake.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Pizzagalli, PhD, Principal Investigator — Mclean Hospital
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts